CLINICAL TRIAL: NCT06360172
Title: The Feasibility of Motivational Interviewing on Emotional Authenticity, Dispositional Optimism, And Academic Motivation Among Nursing Students: A Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3-2024
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Nursing Students
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI (Experimental): Participants in the study group ill obtain six MI sessions. According to Miller and Rollnick's principles, the motivational interviewing group's framework was inspired by the six motivational interviewing sessions in the intervention's booklet Based on the assumption that six to twelve persons in a group are usually necessary for group therapy to be effective, a group of seven students was formed .
  Interventions: Behavioral: Motivational Interviewing
- Control (No Intervention): The control group will receive only the routine teaching with no extra interventions

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational interviewing, or MI, is a collaborative, person-centered counseling technique to uncover and enhance a person's motivation for behavior change
  Arms: MI

SUMMARY:
Motivational interviewing, or MI, is a collaborative, person-centered counseling technique to uncover and enhance a person's motivation for behavior change . MI was first created for the treatment of substance dependence, but it has since been successfully implemented in several fields, including healthcare and education (. Given the vital role that nursing students play in the healthcare system, Saudi Arabia, like many other nations, has realized how important it is to improve the motivation and well-being of its nursing students

DETAILED DESCRIPTION:
This study aims to fill the existing research gap by investigating the feasibility of implementing MI techniques to enhance emotional authenticity, dispositional optimism, and academic motivation among nursing students. By focusing on emotional authenticity, dispositional optimism, and academic motivation among nursing students, the study aims to shed light on the effectiveness of MI techniques in addressing the unique challenges faced by this specific population.

ELIGIBILITY:
Inclusion Criteria:

* Male students to decrease confounding factors, not participating in any type of psychotherapy, and willing to participate in the current study.

Exclusion Criteria:

* Students who complained of any mental disorders or had a previous history of mental problems

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male nursing students
Enrollment: 60 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Kernis-Goldman Authenticity Inventory | 3 months
  The KGAI-3, developed by Kernis and Goldman in 2006, is a 45-item authenticity test of four dimensions. Responses are provided on a 5-point Likert scale, ranging from "Strongly Disagree" to "Strongly Agree"
The Life Orientation Test-Revised form for Adolescents | 3 months
  The original LOT-R is a self-report questionnaire designed to measure dispositional optimism. It was developed by (Scheier, Carver, & Bridges, 1994). The questionnaire consists of ten items: four "filler" items (2, 5, 6, and 8) and three positively formulated things (1, 4, and 10), three negatively formulated items (3, 7, and 9).
Academic Motivation Scale | 3 months
  The Academic Motivation Scale (AMS) is the most popular tool for evaluating academic motivation. (Orsini et al., 2015). A 7-point Likert scale is used to rate each of the 28 items. The self-determination theory, which emphasizes the approach to human motivation and personality, is the theoretical foundation of the AMS

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No